CLINICAL TRIAL: NCT03610477
Title: Effect of Normal Dietary Intake and Medium Chain Triglycerides Supplementation on the Human Microbiome
Brief Title: MiCrobiome dieT Study
Acronym: MCTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1610M95982
Record Dates: First submitted 2018-07-20; First posted 2018-08-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: Microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium Chain Triglyceride (Active Comparator): Participants will be randomized to consume 5% of total energy intake from medium chain triglycerides.
  Interventions: Dietary Supplement: Medium chain triglycerides
- Long Chain Triglyceride (Placebo Comparator): Participants will be randomized to consume 5% of total energy intake from long chain triglycerides.
  Interventions: Dietary Supplement: Long chain triglycerides

INTERVENTIONS:
Dietary Supplement: Medium chain triglycerides — Gel capsules, each containing 1 gram
  Arms: Medium Chain Triglyceride
Dietary Supplement: Long chain triglycerides — Gel capsules, each containing 1 gram
  Arms: Long Chain Triglyceride

SUMMARY:
The human gut microbiome is the community of bacteria that reside within the human intestine. These microbes are constantly exposed to the end-products and partial break-down-products of digestion from the foods consumed each day. Very little is known about the complex interaction of specific dietary components with the microbiome over time in one individual. In order to produce robust analysis of these interactions, longitudinal samples with detailed dietary intake information from healthy human subjects are needed.

The complex relationship between dietary intake and the microbiome, and the potential health implications of human exposure to microbial metabolites, are only beginning to be understood. It is well known that altered dietary intake can trigger rapid, although transient, changes in the composition of the microbiome in as little as 1 to 2 days. The biggest factors in determining microbial response to diet are thought to include an individual's starting microbiome, long-term dietary habits, and environmental exposures.

It is not well understood how small dietary differences from day-to-day impact the microbiome. A longitudinal dataset with accurately recorded dietary data and multiple samples over 17 days will provide valuable insight into the changes that occur at the individual level over time, while controlling for dietary trends and initial microbiome composition.

Medium chain triglycerides (MCTs) have systemic beneficial effects and increase survival in rats by preventing gut injury and permeability following lipopolysaccharide administration, preventing alcohol-induced liver injury, and protecting against the development of colitis in a model of Crohn's disease. Understanding the interaction of MCTs with the microbiome in humans could lead to important advancements in the understanding of how diet impacts the microbiome composition, and ultimately, human health. This proposed study is designed to evaluate the effect of MCTs compared with long chain triglycerides on the normal structure of the microbiome and data will not be used to diagnose, prevent, cure or treat disease.

The purpose of this study is to: 1) investigate the role daily dietary variation plays in microbiome composition and stability, and 2) explore the effect of MCT supplementation on microbiome composition in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult over 18 years

Exclusion Criteria:

* Type 1 diabetes mellitus or insulin dependent type II diabetes mellitus
* Individuals currently maintaining a ketogenic diet
* Women who are currently pregnant or breast feeding
* Use of antibiotics in the last 3 months
* Self-reported pre-existing history of liver disease e.g. cirrhosis or diagnosed fatty liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Microbiome composition | Change from baseline daily for 17 days
  Species-level compositional assessment
Dietary intake variation | Change from baseline daily for 17 days
  Collected as 24-hour daily recalls assessed using novel methods for dietary pattern assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Johnson AJ, Vangay P, Al-Ghalith GA, Hillmann BM, Ward TL, Shields-Cutler RR, Kim AD, Shmagel AK, Syed AN; Personalized Microbiome Class Students; Walter J, Menon R, Koecher K, Knights D. Daily Sampling Reveals Personalized Diet-Microbiome Associations in Humans. Cell Host Microbe. 2019 Jun 12;25(6):789-802.e5. doi: 10.1016/j.chom.2019.05.005. PMID 31194939